CLINICAL TRIAL: NCT00130247
Title: A Prospective Study of Shortening the Duration of Standard Short Course Chemotherapy From 6 Months to 4 Months in HIV-non-infected Patients With Fully Drug-Susceptible, Non-cavitary Pulmonary Tuberculosis With Negative Sputum Cultures After 2 Months of Anti-TB Treatment
Brief Title: Tuberculosis Treatment Shortening Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01-009
Record Dates: First submitted 2005-08-12; First posted 2005-08-15 (Estimated); Results first posted 2010-01-27 (Estimated); Last update posted 2018-11-08 (Actual); Status verified 2010-04-20

CONDITIONS: Tuberculosis
Keywords: Brazil; Philippines; Tuberculosis; Uganda
MeSH Terms: conditions — Tuberculosis | interventions — Ethambutol; Isoniazid; Pyrazinamide; Rifampin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 2EHRZ/2HR arm (Experimental): Daily treatment with isoniazid (INH), rifampicin, ethambutol and pyrazinamide for 2 months followed by 2 months of daily INH plus rifampicin over a maximum time period of 18 weeks.
  Interventions: Drug: Ethambutol; Drug: Isoniazid; Drug: Pyrazinamide; Drug: Rifampin
- 2EHRZ/4HR arm (Active Comparator): Daily treatment with Isoniazid (INH), rifampicin, ethambutol and pyrazinamide for 2 months followed by 4 months of daily INH plus rifampicin over a maximum time period of 28 weeks.
  Interventions: Drug: Ethambutol; Drug: Isoniazid; Drug: Pyrazinamide; Drug: Rifampin

INTERVENTIONS:
Drug: Ethambutol — Mycobacteriostatic agent given to prevent emergence of drug resistance to other 1st line drugs; dosages are 15-25 milligram (mg)/ kilogram (kg)/day (d).
Drug: Isoniazid — Hydrazide of isonicotininc acid; antimicrobial activity is limited to mycobacteria where it inhibits the synthesis of mycolic acids.
Drug: Pyrazinamide — 1st line bactericidal agent; dosages are 15-30 mg/kg/d, up to 2 grams (gm)/d.
Drug: Rifampin — 1st line bactericidal agent which inhibits deoxyribonucleic acid (DNA)-dependent ribonucleic acid (RNA) polymerase; dosages are 10 mg/kg/d (up to 600 mg/d).

SUMMARY:
Tuberculosis (TB) is a serious infection that can affect the lungs and other parts of the body. The usual way to treat TB is to take 4 medicines by mouth every day for 2 months, then take 2 of the same medicines for 4 more months, for a total of 6 months. The purpose of this study is to see if taking 4 months of TB medicines is as effective in curing some TB patients as taking 6 months of TB medicines. Study participants will include 758 human immunodeficiency virus (HIV)-non-infected individuals, ages 18-60. Participants will be treated with 4 standard drugs called isoniazid, rifampicin, pyrazinamide and ethambutol. All individuals will take TB medicines for at least 4 months. After 4 months of treatment, if no TB germs are growing in sputum samples, participants will be assigned to either stop taking TB medicine (4 months of treatment) or to continue taking TB drugs for 2 more months (6 months of treatment). Participants will be involved in study procedures for up to 30 months.

DETAILED DESCRIPTION:
Tuberculosis (TB) is a major global health problem. TB is the current leading cause of death due to an identifiable infectious agent worldwide. One of the highest priorities for tuberculosis control programs is to shorten anti-TB treatment while maintaining its effectiveness. Current 6-month short course chemotherapy regimens are over 95% effective for the treatment of tuberculosis when fully administered. Six months is a long time, however, and patients frequently discontinue anti-TB treatment once their symptoms have improved. The duration of standard short course chemotherapy is one of the major obstacles to its successful application and poses substantial challenges to programs with respect to patient adherence, program resource needs, and logistical requirements for directly observed therapy. The primary objective of this study is to assess the efficacy of shortening anti-TB treatment to 4 months in human immunodeficiency virus (HIV)-non-infected adults with drug-susceptible, non-cavitary pulmonary tuberculosis who convert their sputum culture to negative after 2 months of treatment. Secondary objectives of this study include: comparing pre-treatment sputum bacillary load in patients with and without cavitary disease; compare time after inoculation of BACTEC or Mycobacteria growth indicator tube (MGIT) liquid culture media until positive with semi-quantitative sputum acid fast bacteria (AFB) smear and culture on solid media as measures of pre-treatment sputum bacillary load; and determining the influence of immunologic characteristics of subjects pre-treatment, during treatment and at the end of therapy on rate of bacillary clearance and risk for relapse. A total of 758 HIV-non-infected adults, male or female, 18-60 years of age, with newly diagnosed initial episodes of sputum AFB smear-positive or -negative, culture-positive, non-cavitary, drug-susceptible pulmonary TB who are sputum culture negative after 2 months of anti-TB treatment will be randomly assigned to complete a total of 4 or 6 months of anti-TB therapy. The experimental regimen will include a total of 4 months of anti-TB treatment [2 months of daily isoniazid (INH), rifampicin, pyrazinamide and ethambutol followed by 2 months of daily INH and rifampicin]. The comparative regimen will include a total of 6 months standard short course anti-TB chemotherapy (2 months of daily INH, rifampicin, pyrazinamide and ethambutol followed by 4 months of daily INH and rifampicin). Subjects will be involved in study related procedures for approximately 30 months after beginning the initial anti-TB treatment.

ELIGIBILITY:
Inclusion Criteria:

-Adults, male or female, aged 18-60. -Newly diagnosed initial episodes of pulmonary tuberculosis. Sputum smear-positive and -negative patients are eligible for enrollment. The diagnosis of tuberculosis must be confirmed by culture. Acid fast bacteria (AFB) smear positive patients found later not to have tuberculosis (TB) (i.e. those with non-tuberculous mycobacterial disease) and those without culture confirmation [at least one culture on solid media growing > 10 colonies of Mycobacterium tuberculosis (MTB) or a positive BACTEC or Mycobacteria growth indicator tube (MGIT) enriched liquid culture growing MTB] will be removed from the study. -Chest X-ray and clinical findings consistent with tuberculosis. -Hemoglobin greater than or equal to 8 gm/dL (greater than or equal to 5.0 mmol/L). -Serum creatinine < 2 mg/dL (< 177 micro mol/L). -Serum aspartate aminotransferase (AST) < 1.5 times the upper limit of normal for the testing laboratory, and serum total bilirubin < 1.3 mg/dL (22.2 micro mol/L). -Random serum glucose less than or equal to 150 mg/dl (8.3 mmol/L). -Ambulatory. -Willing to provide informed consent for study participation, provide required specimens for examination, and to undergo and receive results of human immunodeficiency virus (HIV) testing. -Willing to receive supervised anti-TB treatment. -Completion of the required 112 doses of chemotherapy within 18 weeks of starting treatment.

Exclusion Criteria:

-Human immunodeficiency virus (HIV)-infected. -History of prior tuberculosis or history of previous tuberculosis treatment. -Pregnant or breastfeeding. -Cavitary tuberculosis on initial chest X-ray (taken within 14 days of study entry). -Exposure to person(s) with known drug resistant tuberculosis. -Patients receiving chronic steroids or other immunosuppressive medications. -Extra-pulmonary tuberculosis. -Patients with drug resistant tuberculosis (resistance to isoniazid (INH), rifampicin, pyrazinamide or ethambutol). -Professional sex worker, alcoholic and/or intravenous (IV) drug abuser. -Silicosis or other serious chronic medical problems including diabetes mellitus or chronic renal failure. Final determination of eligibility will be made after review of drug susceptibility testing results on an initial sputum isolate and results of all sputum cultures. Pregnant patients may not be enrolled in the study. Patients in the 4 month arm who become pregnant during months 5 and 6 of study participation will be dropped from the study and receive an additional 2 months of treatment with INH and rifampicin.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 394 (Actual)
Dates: Start 2002-04-08 (Actual); Primary Completion 2008-09-02 (Actual); Study Completion 2008-11-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Universidade Federal do Espirito Santo - Duke Hubert-Yeargan Center, Vitória, Espírito Santo, Brazil
- Makati Medical Center, Makati City, National Capital Region, Philippines
- Mulago Hospital Complex, Kampala, Uganda

REFERENCES:
- [Background] Johnson JL, Thiel BA. Time until relapse in tuberculosis treatment trials: implication for phase 3 trial design. Am J Respir Crit Care Med. 2012 Sep 1;186(5):464. doi: 10.1164/ajrccm.186.5.464. No abstract available. PMID 22942350
- [Result] Palaci M, Dietze R, Hadad DJ, Ribeiro FK, Peres RL, Vinhas SA, Maciel EL, do Valle Dettoni V, Horter L, Boom WH, Johnson JL, Eisenach KD. Cavitary disease and quantitative sputum bacillary load in cases of pulmonary tuberculosis. J Clin Microbiol. 2007 Dec;45(12):4064-6. doi: 10.1128/JCM.01780-07. Epub 2007 Oct 10. PMID 17928422
- [Result] Bark CM, Dietze R, Okwera A, Quelapio MI, Thiel BA, Johnson JL. Clinical symptoms and microbiological outcomes in tuberculosis treatment trials. Tuberculosis (Edinb). 2011 Nov;91(6):601-4. doi: 10.1016/j.tube.2011.05.007. Epub 2011 Aug 2. PMID 21813327
- [Result] Colangeli R, Jedrey H, Kim S, Connell R, Ma S, Chippada Venkata UD, Chakravorty S, Gupta A, Sizemore EE, Diem L, Sherman DR, Okwera A, Dietze R, Boom WH, Johnson JL, Mac Kenzie WR, Alland D; DMID 01-009/Tuberculosis Trials Consortium Study 22 Teams. Bacterial Factors That Predict Relapse after Tuberculosis Therapy. N Engl J Med. 2018 Aug 30;379(9):823-833. doi: 10.1056/NEJMoa1715849. PMID 30157391
- [Result] Bark CM, Thiel BA, Johnson JL. Pretreatment time to detection of Mycobacterium tuberculosis in liquid culture is associated with relapse after therapy. J Clin Microbiol. 2012 Feb;50(2):538. doi: 10.1128/JCM.06193-11. Epub 2011 Nov 23. No abstract available. PMID 22116143
- [Result] Johnson JL, Hadad DJ, Dietze R, Maciel EL, Sewali B, Gitta P, Okwera A, Mugerwa RD, Alcaneses MR, Quelapio MI, Tupasi TE, Horter L, Debanne SM, Eisenach KD, Boom WH. Shortening treatment in adults with noncavitary tuberculosis and 2-month culture conversion. Am J Respir Crit Care Med. 2009 Sep 15;180(6):558-63. doi: 10.1164/rccm.200904-0536OC. Epub 2009 Jun 19. PMID 19542476
- [Result] Maciel EL, Brioschi AP, Peres RL, Guidoni LM, Ribeiro FK, Hadad DJ, Vinhas SA, Zandonade E, Palaci M, Dietze R, Johnson JL. Smoking and 2-month culture conversion during anti-tuberculosis treatment. Int J Tuberc Lung Dis. 2013 Feb;17(2):225-8. doi: 10.5588/ijtld.12.0426. PMID 23317958

RESULTS

PARTICIPANT FLOW:
Recruitment Details: HIV-uninfected 18 to 60 year old adults with suspected or newly diagnosed pulmonary tuberculosis were eligible for enrollment at participating sites in Kampala, Uganda; Vitória, Brazil; and Manila/Makati City, the Philippines. Screening began in April 2002 in Uganda, December 2002 in Brazil, and November 2003 in the Philippines.
Pre-assignment Details: Subjects who met eligibility criteria were started on standard chemotherapy and routinely followed during anti-TB therapy. Patients with drug-susceptible TB who were sputum culture negative after 2 months of treatment were randomly assigned at 4 months to stop treatment or received an additional 2 months of daily isoniazid (INH) and rifampicin.
Groups:
- 4-Month Arm: Daily treatment with INH, rifampicin, ethambutol and pyrazinamide for 2 months followed by 2 months of daily INH plus rifampicin over a maximum time period of 18 weeks.
- 6-Month Arm: Daily treatment with INH, rifampicin, ethambutol and pyrazinamide for 2 months followed by 4 months of daily INH plus rifampicin over a maximum time period of 28 weeks.
Period: Overall Study
Arm/Group | 4-Month Arm | 6-Month Arm
Started | 196 | 198
Completed | 194 | 194
Not Completed | 2 | 4
Not completed — Pregnancy | 1 | 0
Not completed — Post-randomization exclusion | 1 | 2
Not completed — Not compliant with DOT | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 4-Month Arm | 6-Month Arm | Total
Number analyzed (Participants) | 196 | 198 | 394
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 196 | 198 | 394
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.2 (10) | 30.3 (10) | 30.8 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 78 | 155
  Male | 119 | 120 | 239
Region of Enrollment [Number; unit: participants]
  Philippines | 47 | 48 | 95
  Brazil | 81 | 81 | 162
  Uganda | 68 | 69 | 137

OUTCOME MEASURES:

1. Primary Outcome: Bacteriologic or Clinical Relapse at 30 Months After Onset of Initial Anti-tuberculosis (TB) Treatment - Intention-to-treat
Description: Patients who presented with TB after completion of study phase treatment but before the end of follow-up were classified as relapses. A bacteriologic relapse was defined as a patient who became consistently culture-positive [defined as at least 1 of the following]: (a) at least 1 sputum mycobacterial culture growing at least 10 colonies of MTB on solid medium; (b) 2 or more respiratory secretion cultures that are positive for MTB in liquid media; or (c) any culture from an extrapulmonary site that is positive for MTB during follow-up after successful completion of initial anti-TB treatment.
Time Frame: 30 months
Population: The intention to treat (ITT) analysis included all 394 fully eligible and randomized patients allocated to the shortened 4-month treatment group (N=196) or the standard 6-month treatment group (N=198). There were no allocated patients excluded in the ITT analysis dataset.
Measure: Number; unit: Participants
Arm/Group | 4-Month Arm | 6-Month Arm
Number analyzed (Participants) | 196 | 198
Participants | 13 | 3
Statistical Analysis 1: Comparison: 4-Month Arm vs 6-Month Arm; Comparison of binomial proportion of relapse: Intention-to-treat; Test type: Non-Inferiority or Equivalence — This two-sided equivalence trial compared the efficacy of 4 and 6 months of treatment. We assumed that the risk of relapse for patients in the 6 month arm was 3.5% and that an absolute difference of 5% (i.e. relapse rate of 8.5%) was clinically meaningful. For a level of significance of 0.05 and 80% power (two sided), we estimated that 284 evaluable subjects per arm were required; Regression, Cox; Risk Difference (RD) = 0.051, 95% CI [0.01 to 0.09] — Confidence interval for difference of binomial proportions adjusted with Hauck Anderson continuity correction

2. Secondary Outcome: Treatment Failures or Relapses at 2 Years After Completion of TB Treatment: Intention to Treat
Description: A culture-positive treatment failure was defined as initial culture conversion but subsequent reversion to culture positivity. A clinical treatment failure was defined as a patient with clinical and/or radiographic evidence of progressive tuberculosis not confirmed by a positive culture after 4 or more months of anti-TB treatment while still receiving treatment. Patients who defaulted before completing study treatment and returned later with culture-positive tuberculosis were termed failures after non-adherence.
Time Frame: 2 years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | 4-Month Arm | 6-Month Arm
Number analyzed (Participants) | 196 | 198
Participants
  Treatment Failures | 0 | 0
  Relapses | 13 | 3

3. Secondary Outcome: Treatment Failures or Relapses at 2 Years After Completion of TB Treatment: Per Protocol
Description: as for outcome 2
Time Frame: 2 years
Population: The per-protocol analysis included all 370 patients (185 per treatment arm) who received the intervention, completed treatment and full follow-up and did not have exogenous reinfection of TB. The 24 excluded subjects included 2 patients with exogenous reinfection of TB, 12 lost to follow-up, 4 deaths, and 6 who did not receive the intervention.
Measure: Number; unit: Participants
Arm/Group | 4-Month Arm | 6-Month Arm
Number analyzed (Participants) | 185 | 185
Participants
  Treatment Failures | 0 | 0
  Relapses | 13 | 3

4. Secondary Outcome: Relapses at 1 and 2 Years
Time Frame: 1 and 2 years after successful completion of initial anti-TB treatment
Population: Analysis includes the 386 patients who received the intervention, completed treatment, and started post-treatment follow-up (193 patients in each treatment arm). Two subjects were lost after completing treatment and contributed no follow-up time, and 6 subjects did not receive the intervention so were not included in the analysis.
Measure: Number; unit: Participants
Arm/Group | 4-Month Arm | 6-Month Arm
Number analyzed (Participants) | 193 | 193
Participants
  Relapses at 1 year | 10 | 3
  Relapses at 2 years | 13 | 3
Statistical Analysis 1: Comparison: 4-Month Arm vs 6-Month Arm; Rate of relapse at 1 year. All patients adherent with treatment and remaining in follow-up at 1 year were included in the calculation of the relapse incidence rate; Test type: Superiority or Other; Regression, Linear; Incidence rate ratio = 3.43, 95% CI [0.94 to 12.5]
Statistical Analysis 2: Comparison: 4-Month Arm vs 6-Month Arm; Rate of relapse at 2 years. All patients adherent with treatment and remaining in follow-up at 2 years were included in the calculation of the relapse incidence rate; Test type: Superiority or Other; Regression, Linear; Incident rate ratio = 4.52, 95% CI [1.29 to 15.9]

5. Secondary Outcome: Acquired Drug Resistance in Patients Who Relapsed
Time Frame: 2 years
Population: This analysis was per protocol and looked for acquired drug resistance among the 13 patients in the 4-Month Arm who relapsed and the 3 patients in the 6-Month Arm who relapsed.
Measure: Number; unit: Participants
Arm/Group | 4-Month Arm | 6-Month Arm
Number analyzed (Participants) | 13 | 3
Participants | 0 | 0

6. Secondary Outcome: Immunologic: Changes in Cytokine Levels in Mycobacterium Tubercolosis (MTB) Antigen-stimulated Whole Blood Culture Supernatants - Results Are Pending
Time Frame: After 2 and 6 months of anti-TB treatment and upon relapse
Reporting Status: Not Posted

7. Secondary Outcome: Immunologic: Store Peripheral Blood Mononuclear Cells (PBMC) - Results Are Pending
Time Frame: Pre-treatment and serum pre-treatment after 2 and 6 months of anti-TB treatment, and at the time of relapse for future immunologic analysis
Reporting Status: Not Posted

8. Secondary Outcome: Immunologic: Changes in Sputum Cytokine Levels - Results Are Pending
Time Frame: After 1 and 2 months of anti-TB treatment
Reporting Status: Not Posted

9. Secondary Outcome: Microbiologic: Changes in Sputum Mycobacterial mRNA - Results Are Pending
Time Frame: At 1 and 2 months of anti-TB treatment, and upon relapse
Reporting Status: Not Posted

10. Primary Outcome: Bacteriologic or Clinical Relapse at 30 Months After Onset of Initial Anti-TB Treatment - Per-protocol
Description: as for outcome 1
Time Frame: 30 months
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | 4-Month Arm | 6-Month Arm
Number analyzed (Participants) | 185 | 185
Participants | 13 | 3
Statistical Analysis 1: Comparison: 4-Month Arm vs 6-Month Arm; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Regression, Cox; Risk Difference (RD) = 0.054, 95% CI [0.01 to 0.10] — Confidence interval for difference of binomial proportions adjusted with Hauck Anderson continuity correction

11. Secondary Outcome: Microbiologic: Time After Inoculation Until Culture Positive in BACTEC 460 or MGIT 960 Enriched Liquid Media After 2 Months in Treatment - Results Are Pending
Time Frame: Months 1, 2, 3, 4, 5, 6, 9, 12, 15, 18, 24, and 30
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 years
Description: Patients reported adverse events at scheduled or unscheduled visits. Adverse event forms were completed by medical officers on site
Arm/Group | 4-Month Arm | 6-Month Arm
Serious Adverse Events (participants affected / at risk) | 19/196 | 22/198
Other Adverse Events (participants affected / at risk) | 170/196 | 164/198
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 4-Month Arm (N=196) | 6-Month Arm (N=198)
Acute Myocardial Infarction (Death) (Cardiac disorders) | 0 (0) | 1 (1)
Bipolar Affective Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Bronchopneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Coronary Arery Occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Cystocele and Perineal Rupture (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Endometrial Polyp (Reproductive system and breast disorders) | 0/77 (0) | 1/78 (1)
Fetal Death (Reproductive system and breast disorders) | 1/77 (1) | 1/78 (1)
Glaucoma in Right Eye (Eye disorders) | 1 (1) | 0 (0)
Gunshot Wound (Abdomen) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gunshot Wound to Head (Death) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Headache (Severe Post-operative) (Nervous system disorders) | 1 (1) | 0 (0)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Hospitalization (Unknown Cause of Abdominal Pain) (Investigations) | 1 (1) | 0 (0)
Hyperhidrosis (General disorders) | 1 (1) | 0 (0)
Malignant Melanoma (Death) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Other Acquired Calcaneus Deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ovarian Cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian Teratoma (Benign) (Reproductive system and breast disorders) | 1/77 (1) | 1/78 (1)
Panuveitis (Eye disorders) | 1 (1) | 0 (0)
Pelvic Abcess (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pre-eclampsia (Reproductive system and breast disorders) | 0/77 (0) | 1/78 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 10/77 (10) | 13/78 (14)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Suffocation (Death) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Surgical Intervention on Right Shoulder (Surgical and medical procedures) | 0 (0) | 1 (1)
Tracheal Plastic Repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Uterine Myoma (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vocal Cord Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4-Month Arm (N=196) | 6-Month Arm (N=198)
Abdominal Pain (Gastrointestinal disorders) | 48 (63) | 49 (59)
Acne (Skin and subcutaneous tissue disorders) | 14 (15) | 16 (17)
Appetite Lost (Metabolism and nutrition disorders) | 39 (49) | 30 (35)
Arthralgia (Musculoskeletal and connective tissue disorders) | 64 (92) | 64 (87)
Back Pain (Musculoskeletal and connective tissue disorders) | 34 (46) | 31 (36)
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 70 (115) | 52 (77)
Coryza (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 10 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 104 (186) | 90 (162)
Diarrhea (Gastrointestinal disorders) | 15 (20) | 10 (10)
Dizziness (Nervous system disorders) | 18 (20) | 17 (18)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 17 (18) | 9 (9)
Fever (General disorders) | 87 (148) | 67 (103)
Flu (Infections and infestations) | 40 (63) | 27 (46)
Headache (Nervous system disorders) | 64 (102) | 46 (66)
Hemoptysis (Blood and lymphatic system disorders) | 15 (19) | 15 (19)
Insomnia (Psychiatric disorders) | 8 (11) | 11 (15)
Malaise (General disorders) | 17 (22) | 15 (18)
Malaria (Infections and infestations) | 9 (12) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 15 (16)
Nausea (Gastrointestinal disorders) | 20 (31) | 32 (41)
Pain in Limb (Musculoskeletal and connective tissue disorders) | 6 (8) | 11 (14)
Produce Sputum (Respiratory, thoracic and mediastinal disorders) | 48 (57) | 39 (50)
Pruritis (Skin and subcutaneous tissue disorders) | 46 (57) | 43 (52)
Purulent Sputum (Respiratory, thoracic and mediastinal disorders) | 34 (40) | 27 (33)
Rash (Skin and subcutaneous tissue disorders) | 18 (20) | 15 (15)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 12 (17) | 17 (19)
Rigors (General disorders) | 13 (15) | 12 (15)
Skin Lesion (Skin and subcutaneous tissue disorders) | 15 (21) | 9 (22)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 14 (15) | 10 (10)
Sweating (General disorders) | 13 (15) | 17 (22)
Tinea Infection (Infections and infestations) | 10 (12) | 6 (9)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 33 (50) | 27 (39)
Vomiting (Gastrointestinal disorders) | 15 (18) | 16 (19)
Weight Loss (Metabolism and nutrition disorders) | 24 (29) | 20 (26)

LIMITATIONS AND CAVEATS:
Enrollment was stopped early and the number of patients enrolled was 1/2 of the original sample size. The study was completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No